CLINICAL TRIAL: NCT00835926
Title: Safety and Immunogenicity of Influenza Virus Vaccine USP Trivalent Types A and B (Zonal Purified Subvirion) Fluzone® 2003/2004
Brief Title: A Study to Evaluate the Safety and Immune Responses to Fluzone® Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC16
Record Dates: First submitted 2009-01-27; First posted 2009-02-04 (Estimated); Results first posted 2009-10-26 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza; Fluzone®
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluzone® Vaccine Group 1 (Experimental): Participants aged 18 to 59 years at enrollment - Fluzone® Group
  Interventions: Biological: Influenza virus vaccine
- Fluzone® Vaccine Group 2 (Experimental): Participants aged 60 years and older at enrollment - Fluzone® Group
  Interventions: Biological: Influenza virus vaccine

INTERVENTIONS:
Biological: Influenza virus vaccine — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Fluzone® Vaccine Group 1
Biological: Influenza virus vaccine — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Fluzone® Vaccine Group 2

SUMMARY:
To describe the safety during days 0 to 21 following injection of the 2003-2004 formulation of the inactivated, split-virion influenza vaccine Fluzone® in subjects aged 18-59 years and subjects aged ≥ 60 years.

To describe the immune response at 21 days following injection of the 2003-2004 formulation of the inactivated, split-virion influenza vaccine Fluzone®, in subjects aged 18-59 years and subjects aged ≥ 60 years.

DETAILED DESCRIPTION:
Safety will be assessed throughout the trial period. Using antigens provided by Aventis Pasteur Inc., pre- and post-vaccination serum antibody titers for each of the three vaccine strains will be measured.

ELIGIBILITY:
Inclusion Criteria :

* Age of 18 years or greater.
* Ambulatory.
* In reasonably good health as assessed by the investigator.
* Available for duration of the study (21 days + 2d).
* Willing and able to meet protocol requirements.
* Willing and able to give informed consent.

Exclusion Criteria :

* Self-reported allergy to egg proteins, chicken proteins, or one of the constituents of the vaccine, such as thimerosal or formaldehyde.
* An acute illness with or without fever (temperature >100.4°F) in the 72 hours preceding enrollment in the trial.
* Clinically significant findings in vital signs (including temperature >100.4°F) or review of systems.
* Self-reported history of severe adverse event to any influenza vaccine.
* Vaccination against influenza in the 6 months preceding enrollment in the study.
* Any vaccination in the 14 days preceding enrollment in the study or scheduled between Visit 1 and Visit 3.
* Participation in any other experimental drug or vaccine trial within the 30 days preceding enrollment into the study.
* Immunosuppressive therapy including long-term (> 2 weeks) systemic corticosteroids or cancer therapy within the past 3 months or ongoing.
* Receipt of blood or blood products within the 3 months preceding enrollment in the study.
* Diabetes
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine (e.g., existing severe chronic illness such as pulmonary disorders, cardiovascular disorders, chronic blood disorders, etc.).
* Person deprived of freedom by an administrative or court order (having legal or medical guardian).
* For women of childbearing age, a positive urine pregnancy test, breast feeding, or not using a medically approved and reliable form of contraception (oral contraceptives or double barrier method) for the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2003-07; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 25 July 2003 to 26 August 2003 at 1 US site.
Pre-assignment Details: A total of 121 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Fluzone® Vaccine Group 1: Participants were 18 to 59 years old at enrollment in the study
- Fluzone® Vaccine Group 2: Participants were 60 years or older at enrollment in the study
Period: Overall Study
Arm/Group | Fluzone® Vaccine Group 1 | Fluzone® Vaccine Group 2
Started | 61 | 60
Completed | 61 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone® Vaccine Group 1 | Fluzone® Vaccine Group 2 | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 60 | 5 | 65
  >=65 years | 0 | 55 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 40.7 (10.43) | 73.7 (6.16) | 57.1 (18.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 39 | 87
  Male | 13 | 21 | 34
Region of Enrollment [Number; unit: participants]
  United States | 61 | 60 | 121

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection Site and Systemic Reactions Post-Vaccination With Fluzone®
Description: Solicited injection site reactions: Erythema, bruising, induration, and Pain at injection site.
  Solicited systemic reaction: Fever (temperature), chills, rash, headache, cough, runny nose, nausea, vomiting, diarrhea, malaise, myalgia, and arthralgia
Time Frame: Days 0 to 3 Post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants, intent-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone® Vaccine Group 1 | Fluzone® Vaccine Group 2
Number analyzed (Participants) | 61 | 60
Percentage of Participants
  Any Erythema | 15 | 7
  Grade 3 Erythema (> 5 cm) | 0 | 2
  Any Induration | 20 | 12
  Grade 3 Induration (> 5 cm) | 2 | 0
  Any Bruising | 10 | 3
  Grade 3 Bruising (> 5 cm) | 0 | 2
  Any Pain | 75 | 12
  Grade 3 Pain (Decreased ability to move arm) | 0 | 0
  Any Fever | 0 | 2
  Grade 3 Fever (Incapacitating) | 0 | 0
  Any Chills | 5 | 2
  Grade 3 Chills (Incapacitating) | 0 | 0
  Any Rash | 0 | 0
  Grade 3 Rash (Incapacitating) | 0 | 0
  Any Headache | 23 | 7
  Grade 3 Headache (Incapacitating) | 2 | 2
  Any Cough | 0 | 2
  Grade 3 Cough (Incapacitating) | 0 | 0
  Any Runny Nose | 5 | 3
  Grade 3 Runny Nose (Incapacitating) | 0 | 0
  Any Nausea | 7 | 0
  Grade 3 Nausea (Incapacitating) | 0 | 0
  Any Vomiting | 2 | 0
  Grade 3 Vomiting (Incapacitating) | 0 | 0
  Any Diarrhea | 3 | 0
  Grade 3 Diarrhea (Incapacitating) | 0 | 0
  Any Malaise | 10 | 3
  Grade 3 Malaise (Incapacitating) | 2 | 2
  Any Myalgia | 13 | 5
  Grade 3 Myalgia (Incapacitating) | 0 | 0
  Any Arthralgia | 5 | 3
  Grade 3 Arthralgia (Incapacitating) | 0 | 0

2. Primary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition Antibodies Before and After Vaccination With Fluzone®
Description: Hemagglutination inhibition antibodies is a measure of the serum antibody to the influenza virus in the vaccine as determined by the hemagglutinin inhibition (HAI) assay.
Time Frame: Day 0 and Day 21 Post-vaccination
Population: The Geometric mean titers were analyzed in the per-protocol immunogenicity population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone® Vaccine Group 1 | Fluzone® Vaccine Group 2
Number analyzed (Participants) | 61 | 60
Titers
  A/Panama/2007/99 Pre-Dose | 29.6 [22.6 to 38.7] | 20.4 [15.9 to 26.2]
  A/Panama/2007/99 Post-Dose | 67.1 [50.7 to 88.7] | 37.5 [29.5 to 47.7]
  A/New Caledonia/20/99 Pre-Dose | 18.3 [13.6 to 24.7] | 9.5 [7.7 to 11.6]
  A/New Caledonia/20/99 Post-Dose | 46.3 [34.3 to 62.5] | 15.1 [12.1 to 18.9]
  B/Hong Kong/1434/2002 Pre-Dose | 10.7 [8.6 to 13.3] | 8.2 [6.8 to 9.7]
  B/Hong Kong/1434/2002 Post-Dose | 27.8 [22.1 to 34.9] | 15.9 [12.6 to 20.1]

3. Primary Outcome: Percentage of Participants With a ≥ 4-Fold Rise in Serum Hemagglutination Inhibition Antibody Titers Post-Vaccination With Fluzone®
Description: as for outcome 2
Time Frame: Day 21 Post-vaccination
Population: The vaccine antibody fold rise analysis was in the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone® Vaccine Group 1 | Fluzone® Vaccine Group 2
Number analyzed (Participants) | 61 | 60
Percentage of Participants
  A/Panama/2007/99 | 28 | 18
  A/New Caledonia/20/99 | 30 | 8
  B/Hong Kong/1434/2002 | 38 | 22

4. Primary Outcome: Percentage of Participants With Serum Hemagglutination Inhibition Antibody Titers ≥ 40 Post-Vaccination With Fluzone®
Description: as for outcome 2
Time Frame: Day 21 Post-vaccination
Population: The Fluzone® antibody titers were analyzed in the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone® Vaccine Group 1 | Fluzone® Vaccine Group 2
Number analyzed (Participants) | 61 | 60
Percentage of Participants
  A/Panama/2007/99 | 74 | 60
  A/New Caledonia/20/99 | 62 | 25
  B/Hong Kong/1434/2002 | 41 | 25

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Fluzone® Vaccine Group 1 | Fluzone® Vaccine Group 2
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 8/61 | 2/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone® Vaccine Group 1 (N=61) | Fluzone® Vaccine Group 2 (N=60)
Headache (Nervous system disorders) | 8 (12) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications